CLINICAL TRIAL: NCT03087500
Title: Physiologic Biomarkers Within the Functional Spectrum of Down Syndrome
Brief Title: Physiological Abnormalities Associated with Down Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Funding fell through
Sponsor: University of Arkansas (Other)
Collaborators: Down Syndrome Research Foundation (Unknown); Arkansas Children Research Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 206522
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2017-10

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Typically Developing Participants; Children; Adolescents; Adults
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Biomarkers of oxidative stress (GSH/GSSG)
  * Biomarkers of reduced methylation capacity (SAM/SAH)
  * Biomarkers of mitochondrial energetics
  * Metabolomics (Urine, Blood)
  * Salivary inflammatory cytokines (IL-1, IL2, IL-6, TNFα)
  * DNA methylation array (epigenetic profile); total DNA methylation
  * Folate Receptor Autoantibody (Blocking and Binding)
  * Thyroid Function (Thyroid Stimulating Hormone, T3, Reverse T3 and free and total T4)
  * Microbiome Analysis (Stool)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Down Syndrome (DS): 120 clinically confirmed full trisomy 21, age 3-50 years of both sexes will be recruited as the target study population. Half of the individuals (n=60) will be children (3-17 years of age) while half (n=60) will be adults (18-50 years of age)
  Interventions: Other: There is no other intervention, only clinical treatment.
- Typically Developing Controls: 60 typically developing individuals age 3-50, age and gender matched to at least one participant with DS. Half of the controls (n=30) will be age and gender match to children with DS and half (n=30) will be age and gender matched to adults with DS.
  Interventions: Other: There is no other intervention, only clinical treatment.

INTERVENTIONS:
Other: There is no other intervention, only clinical treatment. — There is no other intervention, only clinical treatment.

SUMMARY:
The overall goal of this study is to evaluate biomarkers of oxidative stress, mitochondrial function, and DNA methylation (epigenetics) in order to determine the extent to which these biomarkers are related to cognitive, behavioral and adaptive function in Down Syndrome. The inter-relationship between measurable biomarkers and functional/cognitive abilities will move beyond genetics to provide unprecedented new knowledge and a broader understanding of the underlying pathophysiology and abnormal gene expression induced by trisomy 21.

DETAILED DESCRIPTION:
The Investigators preliminary evidence indicates that people with DS have metabolic biomarkers associated with oxidative stress (GSH/GSSG) and reduced methylation capacity (SAM/SAH) as well as abnormal DNA methylation (epigenetics). The investigative team hypothesize that these abnormal metabolic processes contribute to abnormalities in behavior and development associated with trisomy 21; this connection has never been investigated. Confirming and expanding on the preliminary data would provide new understanding of the biological and functional etiology of the behavioral and developmental delays associated with Trisomy 21. Further, establishing the underlying relationship between metabolic abnormalities and behavioral/cognitive function over the age spectrum can provide strong support for the design of future treatments of individuals with DS aimed at improving their behavior and development. In addition, these biomarkers may also prove to be predictive biomarkers for the risk of developing ASD like behaviors or Alzheimer's disease in this population. Finally, examining the modulating role of diet in the severity of biological abnormalities will provide new information for lifestyle guidance to improve biomarkers and potentially minimize the medical co-morbidities associated with trisomy 21.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or guardian ability to consent/assent and willing to comply with protocol requirements

Exclusion Criteria:

1. Trisomy translocation or mosaics.
2. Untreated hypothyroidism
3. Known history of liver disease, renal disease, Hepatitis B or C or HIV
4. Recent infection with fever or requiring hospitalization within past 30 days.
5. Any medical condition, use of medications, nutrient or herbal supplements that would interfere with the study results as determined by the PI
6. Chemotherapy
7. Recent surgery (within 2 months)
8. Untreated Epilepsy
9. Any chronic medical/behavioral condition and/or treatments that may interfere with study related outcomes, as determined by PI
10. Dementia
11. History of a significant adverse reaction to a prior blood draw
12. Any other historical event/information that may, in the opinion of the PI, be a reason to exclude the child from participation.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Downs Syndrome: 120 clinically confirmed full trisomy 21, age 3-50 years of both sexes will be recruited as the target study population. Half of the individuals (n=60) will be children (3-17 years of age) while half (n=60) will be adults (18-50 years of age) Control Subjects: 60 typically developing individuals age 3-50, age and gender matched to at least one participant with DS. Half of the controls (n=30) will be age and gender match to children with DS and half (n=30) will be age and gender matched to adults with DS.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Microbiome Analysis | 2 years
  Stool will be collected for Microbiome Analysis on cases and controls
Mitochondrial Function Analysis | 2 years
  The Seahorse XR extracellular flux analyzer will be used to measure mitochondrial function in cases and controls
Oxidative Stress Analysis | 2 years
  Thiol measurements will be collected and analyzed between cases and controls
Immune Function | 2 years
  Salivary measurements of cytokines will be collected on cases and controls
Metabolomics | 2 years
  Urine will be collected for metabolomics analysis on cases and controls
Epigenetics | 2 years
  Epigenetics will be evaluated on cases and controls
Folate Receptor Alpha Autoantibody (FRAA) | 2 years
  Serum will be collected for FRAA analysis on cases and controls
Thyroid Function | 2 years
  Thyroid measures of Thyroid Stimulating Hormone (TSH), T3, Reverse T3 and free and total T4 will be evaluated on cases and controls
Diet | 2 years
  Examine the modulating role of diet in the severity of biological abnormalities will provide new information for lifestyle guidance to improve biomarkers and potentially minimize the medical co-morbidities associated with trisomy 21. Dietary contributions will be evaluated on cases and controls

CONTACTS AND LOCATIONS:
Overall Officials: Richard Frye, Principal Investigator — Arkansas Childrens Research Institute

IPD SHARING:
Plan to Share IPD: No